CLINICAL TRIAL: NCT06934590
Title: An Open-label, Dose Escalation, Phase I Study to Evaluate Safety and Tolerability of RX001 in Patients With KRAS Mutant Advanced Non-small Cell Lung Cancer
Brief Title: Evaluate Safety and Tolerability of RX001 in Patients With KRAS Mutant Advanced NSCLC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GeneCraft Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-LCP1001
Record Dates: First submitted 2025-04-02; First posted 2025-04-18 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: KRAS; NSCLC; RUNX3; AAV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RX001 (Experimental): RX001
  Interventions: Drug: RX001

INTERVENTIONS:
Drug: RX001 — Subjects will receive a single RX001 (AAV-hRUNX3) treatment via Intra-tumoral injection

SUMMARY:
This is an open-label, dose-escalation Phase I study to evaluate the safety and tolerability of RX001 monotherapy in patients with advanced KRAS mutant NSCLC. Subjects aged ≥19 years with advanced NSCLC with KRAS mutations will be enrolled. Based on the investigator's judgment of the lung tumor location, RX001 will be administered as a single intratumoral treatment via bronchoscopy or CT-guided percutaneous injection. Additionally, after conducting safety, tolerability, and preliminary anti-tumor efficacy assessments for all subjects up to Week 12 (D84) following IP administration, the collected data will be reviewed by the SRC for a comprehensive evaluation. If the IP is designated for long-term follow-up studies, monitoring for malignant tumor formation and other SAEs specified by the Ministry of Food and Drug Safety (MFDS) will be conducted for a minimum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥19 years, male or female
* Subject with histologically and/or cytologically confirmed, unresectable advanced NSCLC for radical cure that are confirmed as PD for the standard of care currently known to have clinical benefits, or for which no currently available standard of care exists due to intolerance, ineligibility, treatment refusal, etc.
* Subjects must have at least one evaluable and injectable lesion as assessed on CT images based on RECIST version 1.1.
* Subjects with valid biopsy results documented the presence of KRAS mutation.
* Subjects with an ECOG performance status of 0 or 1 and an expected survival of at least 12 weeks at the time of study participation.
* Subjects with adequate hematologic and terminal organ function.
* Subjects must voluntarily sign an informed consent form approved by the IRB. Subjects must have the willingness and ability to comply with all procedures required by the protocol.

Exclusion Criteria:

* Subjects must not meet any of the following conditions:
* Subjects with a history of or current comorbidities including:

  1. Hematologic malignancies, such as lymphoma, or any other malignant tumors apart from the indication of this study.
  2. Subjects with the cardiovascular conditions such as unstable angina and/or myocardial infarction within 1 year prior to screening
  3. Subjects with the pulmonary baseline conditions:
  4. Blood coagulation disorder
  5. Active bleeding disorders (including gastrointestinal bleeding)
* Subjects who have received antithrombotics, including antiplatelets or anticoagulants
* Subjects who have received anticancer therapies within 28 days prior to trial participation, or who have not recovered or stabilized from all AEs caused by such treatments to baseline levels
* Subjects who have received radical radiotherapy within 6 weeks prior to trial participation etc.
* Subjects who have received live vaccines or attenuated vaccines within 4 weeks prior to study participation
* Subjects with active HBV or HCV, or HIV positive
* Subjects with severe infections requiring antibiotics, antifungal agents, or antiviral agents, or those with uncontrolled active infectious diseases
* Subjects with any form of primary immunodeficiency or active autoimmune diseases
* Subjects who have previously received intratumoral therapy for the target lesion
* Ineligibility or inability to participate in the study at the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related serious adverse event (SAE) rate | Observation for 12 weeks following a single dose
  Incidence of SAEs throughout the study
  SAE: an adverse event or suspected adverse reaction is considered "serious" if, in the view of the investigator, it results in any of the following outcomes:
  Death or a life-threatening adverse event Inpatient hospitalization or prolongation of existing hospitalization A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions A congenital anomaly/birth defect Any other important medical event that does not fit the criteria above but, based upon appropriate medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above

SECONDARY OUTCOMES:
Objective response rate (ORR) | Observation for 12 weeks following a single dose
  * ORR = percentage of participants with complete response + partial response.
  * Complete response (CR): Disappearance of all target lesions.
  * Partial response (PR): At least a 30% decrease in the diameters of target lesions, taking as reference the baseline diameters.
Progression-free survival (PFS) | Observation for 12 weeks following a single dose
  PFS is defined as the time from date of treatment initiation to disease progression or death from any cause, whichever occurs first.
Target Tumor Size | Observation for 12 weeks following a single dose
  Changes in the maximum length of the target lesion

OTHER OUTCOMES:
Immune response assessment | Observation for 12 weeks following a single dose
  Evaluate the formation of anti-AAV2 antibodies
Viral Shedding Profile Assessment | Observation for 12 weeks following a single dose
  Assess the extent of vector DNA shedding in saliva, urine, feces, and other excreta following administration

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The current position is "No" due to pending internal policy decisions. However, revision of internal regulations is under review to allow for potential future data sharing and registry compliance.